CLINICAL TRIAL: NCT02206035
Title: Phase II Open-Label Trial of Tacrolimus/Methotrexate and Tocilizumab for the Prevention of Acute Graft-Versus-Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Study of Tacrolimus/Methotrexate and Tocilizumab to Prevent Acute Graft-Versus-Host Disease (AGVD) After Allogeneic Hematopoietic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William R. Drobyski, MD (Other)
Responsible Party: Sponsor-Investigator, William R. Drobyski, MD, Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00023000
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Tacrolimus; Methotrexate; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) (Experimental): Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant. Methotrexate will be dosed at 15 mg/m2 Day +1 and 10mg/m2 Days +3, +6 and +11. Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1
  Interventions: Drug: Tacrolimus; Drug: Methotrexate; Drug: Tocilizumab

INTERVENTIONS:
Drug: Tacrolimus — Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant.
  Other Names: fujimycin; FK506
Drug: Methotrexate — Methotrexate will be dosed at 15 mg/m2 Day +1 and 10mg/m^2 Days +3, +6 and +11.
  Other Names: Trexall
Drug: Tocilizumab — Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1.
  Other Names: Actemra

SUMMARY:
This is a phase II open label trial designed to evaluate the efficacy of Tac/MTX/Toc in preventing graft versus host disease (GVHD). Outcomes of patients on this clinical trial will be compared to those of contemporary controls from the CIBMTR.

DETAILED DESCRIPTION:
This is a Phase II open label trial designed to evaluate the efficacy of Tacrolimus (Tac), Methotrexate (MTX) and Tocilizumab (Toc) (combined Tac/MTX/Toc) in preventing graft versus host disease (GVHD) after allogeneic hematopoietic stem cell transplantation compared to a contemporary control cohort selected from the Center for International Bone Marrow Transplant Research (CIBMTR) that is treated with standard methotrexate and tacrolimus for GVHD prevention. The control group of patients will satisfy similar eligibility requirements as the patients enrolled in the clinical trial and they will be matched for relevant clinical variables (age, sex, conditioning regimen, disease, graft source, etc).

Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 post transplant. Methotrexate will be dosed at 15 mg/m^2 Day +1 and 10mg/m^2 Days +3, +6 and +11. Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1.

Ancillary Study:

The ancillary study will evaluate whether tocilizumab is effective at positively impacting mood, fatigue, sleep, and pain in a group of individuals undergoing allogeneic hematopoietic stem cell transplantation as compared to individuals not receiving tocilizumab. We will also assess whether tocilizumab alters gene expression and Rap1 prenylation in a manner that may reduce further progression or relapse of cancer after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with acute leukemia, chronic myelogenous leukemia, myeloproliferative disease and myelodysplasia with less than 5% of blasts in the bone marrow
3. Patients with chronic lymphocytic leukemia/small lymphocytic lymphoma, Non-Hodgkin Lymphoma or Hodgkin Disease with chemosensitive disease at time of transplant
4. Planned conditioning regimens including combination of busulfan and fludarabine or busulfan and cyclophosphamide
5. Transplantation with T-cell-replete grafts
6. Bone marrow or mobilized peripheral blood cell grafts
7. Patients must have either a sibling donor (6/6 match at human leukocyte antigens (HLA-A, -B and -DRB1) or a unrelated donor (8/8 match at HLA-A, -B, -C and -DRB1)
8. Cardiac function: Ejection fraction at rest >45% for myeloablative conditioning or >40% for reduced intensity conditioning
9. Estimated creatinine clearance greater than 50 mL/minute (using the Cockcroft-Gault formula and actual body weight)
10. Pulmonary function: Diffusing Capacity of Lung for Carbon Monoxide (DLCO) ≥40% (adjusted for hemoglobin) and FEV1≥50%
11. Liver function: total bilirubin < 1.5 x the upper limit of normal and alanine aminotransferase (ALT) / aspartate aminotransferase (AST) < 2.5x the upper normal limit
12. Signed informed consent

Exclusion Criteria:

1. Prior allogeneic hematopoietic cell transplant (HCT)
2. Karnofsky Performance Score <70%
3. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression of infectious disease or no clinical improvement) at time of enrollment
4. Prior intolerance or allergy to Tocilizumab
5. Use of rituximab, alemtuzumab, anti-thymocyte globulin (ATG) or other monoclonal antibody at time of conditioning regimen
6. History of diverticulitis, Crohn's disease or ulcerative colitis
7. History of demyelinating disorder
8. Pregnant and lactating women
9. Patients with a history of rheumatologic disorders who have previously received Tocilizumab

Eligibility for the Control Arm

Patients in the control arm will be identified from patients reported to the CIBMTR from U.S centers. Control patients will be required to satisfy similar eligibility requirements as patients being enrolled in the clinical trial. Patients will need to fulfill the same inclusion criteria for the clinical trial according to Section 2.4.1, plus the following:

1. Receive Tac/MTX as the sole GVHD prophylaxis approach
2. Receive the same regimens as specified in Table 2.5
3. Year of transplant from 2010 to 2013

Exclusion criteria for the controls:

1. Karnofsky Performance Score < 70%

Data for all eligible patients will be used to constitute the control database for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Drobyski, MD, Principal Investigator — Medical College of Wisconsin; Marcelo Pasquini, MD, Principal Investigator — Medical College of Wisconsin; Jennifer Knight, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson D, O'Hara MW, Simms LJ, Kotov R, Chmielewski M, McDade-Montez EA, Gamez W, Stuart S. Development and validation of the Inventory of Depression and Anxiety Symptoms (IDAS). Psychol Assess. 2007 Sep;19(3):253-68. doi: 10.1037/1040-3590.19.3.253. PMID 17845118
- [Background] D'Souza A, Lee S, Zhu X, Pasquini M. Current Use and Trends in Hematopoietic Cell Transplantation in the United States. Biol Blood Marrow Transplant. 2017 Sep;23(9):1417-1421. doi: 10.1016/j.bbmt.2017.05.035. Epub 2017 Jun 9. PMID 28606646
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The populations used for historical controls were not recruited by theses investigators. To obtain matched controls, the number of records analyzed exceeds the number recruited locally for the interventional arm.
  This investigation was conducted jointly by two research teams investigating the clinical effects, and the other investigating behavioral effects.. Each investigational team selected a population of matched historic controls appropriate to its outcome measures.
Groups:
- Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc): Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant. Methotrexate will be dosed at 15 mg/m^2 Day +1 and 10mg/m^2 Days +3, +6 and +11. Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1
  Tacrolimus: Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant.
  Methotrexate: Methotrexate will be dosed at 15 mg/m^2 Day +1 and 10mg/m^2 Days +3, +6 and +11.
  Tocilizumab: Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1.
- Historical Control Arm (Primary Outcome Measure): This population was derived from case reports to the Center for International Blood and Marrow Transplant Research® (Milwaukee, WI) comprising patients receiving a first allogeneic transplant at a US site excluding the Medical College of Wisconsin. Additional population details can be found in D'Souza, 2017. (n=130)
  Race and ethnicity information was not collected for this control population.
- Historical Control Arm (Secondary Outcome Measures): This population was derived from case reports from individuals participating in a longitudinal study evaluating biobehavioral effects on recovery following allogeneic hematopoietic cell transplantation at the University of Wisconsin-Madison. Patients received prophylaxis for graft versus host disease with methotrexate/tacrolimus. No patients received tocilizumab. (n=204). Patients receiving a second transplant; BCNU/carmustine, etoposide, cytarabine, and melphalan (BEAM) conditioning; total body irradiation; anti-thymocyte globulin, sirolimus; cord blood transplant; or cyclosporine/mycophenolate mofetil prophylaxis for graft versus host disease were excluded. Results presented are further limited to patients with acute myelogenous leukemia, acute lymphocytic leukemia, chronic myelogenous leukemia, and myelodysplastic syndrome to match the treatment population (n = 29).
Period: Overall Study
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Started | 45 | 130 | 204
Completed | 35 | 130 | 29
Not Completed | 10 | 0 | 175
Not completed — Physician Decision | 10 | 0 | 175

BASELINE CHARACTERISTICS:
Groups:
- Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc): Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant. Methotrexate will be dosed at 15 mg/m2 Day +1 and 10mg/m^2 Days +3, +6 and +11. Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1
  Tacrolimus: Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant.
  Methotrexate: Methotrexate will be dosed at 15 mg/m^2 Day +1 and 10mg/m^2 Days +3, +6 and +11.
  Tocilizumab: Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1.
- Historical Control Arm (Secondary Outcome Measures): This population was derived from case reports from individuals participating in a longitudinal study evaluating biobehavioral effects on recovery following allogeneic hematopoietic cell transplantation at the University of Wisconsin-Madison. Patients received prophylaxis for graft versus host disease with methotrexate/tacrolimus. No patients received tocilizumab. (n=204). Patients receiving a second transplant; BCNU/carmustine, etoposide, cytarabine, and melphalan (BEAM) conditioning; total body irradiation; anti-thymocyte globulin; sirolimus; cord blood transplant; or cyclosporine/mycophenolate mofetil prophylaxis were excluded. Results presented are further limited to patients with acute myelogenous leukemia, acute lymphocytic leukemia, chronic myelogenous leukemia, and myelodysplastic syndrome to match the treatment population (n = 29).
- Total: Total of all reporting groups
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures) | Total
Number analyzed (Participants) | 35 | 130 | 29 | 194
Age, Continuous [Median (Full Range); unit: years] | 66 [22 to 76] | 64 [23 to 74] | 54 [44 to 64] | 62 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender demographics was not collected for the Historical Control Arm (Primary Outcome Measure) population.
  Participants
    Known Gender: number analyzed (Participants) | 35 | 0 | 29 | 64
    Known Gender: Female | 13 |  | 9 | 22
    Known Gender: Male | 22 |  | 20 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 28 | 28
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 0 | 0 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 130 | 0 | 140
Region of Enrollment [Number; unit: participants]
  United States | 35 | 130 | 29 | 194

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Not Experiencing Grade II-IV Acute Graph Versus Host Disease (aGVHD)
Description: This measure is the number of subjects who did not experience grade II-IV aGVHD at or before day 180 comparing recipients of tacrolimus (Tac), methotrexate (MTX), and tocilizumab (Toc) to a contemporary control population abstracted from a database maintained by the Center for International Blood and Marrow Transplant Research (CIBMTR). The staging of aGVHD was according to the criteria of Przepiorka, et al., 1995 which assigns a score to the clinical status of multiple organ systems aggregated to determine the clinical stage. A higher stage indicates more severe aGVHD symptoms and poorer clinical outcome.
Time Frame: Day 180
Population: The Historical Control Arm (Secondary Outcome Measures) cohort was included in this study for comparison of the behavioral results (Outcome Measures 2-6). The occurrence of aGVHD was not collected for this population. The Historical Control Arm (Secondary Outcome Measures) cohort has no clinical outcome for comparison and is not included in the analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Historical Control Arm (Primary Outcome Measure): This population was derived from case reports to the Center for International Blood and Marrow Transplant Research® (Milwaukee, WI) comprising patients receiving a first allogeneic transplant at a US site excluding the Medical College of Wisconsin. Additional population details can be found in D'Souza, 2017.05.035. (n=130)
  Race and ethnicity information was not collected for this control population.
- Historical Control Arm (Secondary Outcome Measures): This population was derived from case reports from individuals participating in a longitudinal study evaluating biobehavioral effects on recovery following allogeneic hematopoietic cell transplantation at the University of Wisconsin-Madison. Patients received prophylaxis for graft versus host disease with methotrexate/tacrolimus. No patients received tocilizumab. (n=204). Patients receiving a second transplant, BEAM conditioning (BCNU/carmustine, etoposide, cytarabine, and melphalan), total body irradiation, anti-thymocyte globulin, sirolimus, cord blood transplant, or cyclosporine/mycophenolate mofetil GVHD prophylaxis were excluded. Results presented are further limited to patients with acute myelogenous leukemia, acute lymphocytic leukemia, chronic myelogenous leukemia, and myelodysplastic syndrome to match the treatment population (n = 29).
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Number analyzed (Participants) | 35 | 130 | 0
Participants | 3 | 18 | 0

2. Secondary Outcome: Score of Depressive Symptoms Using General Depressive Subscale of the Inventory of Depression and Anxiety Symptoms (IDAS) Instrument
Description: The measure of depressive symptoms will be determined from the Inventory of Depression and Anxiety Symptoms (IDAS) instrument. The IDAS contains 10 specific symptom scales: Suicidality, Lassitude, Insomnia, Appetite Loss, Appetite Gain, Ill Temper, Well-Being, Panic, Social Anxiety, and Traumatic Intrusions (see Watson, 2007). The General Depression subscale of the IDAS and includes a subset of 20 five-item Likert-style questions (1= "Not at All" to 5-= "Extremely") with a scoring range of 20-100. Higher scores indicate more severe symptoms.
Time Frame: Baseline, Day 28, Day 100 and Day 180
Population: The Historical Control Arm (Primary Outcome Measure) cohort was included in this study for comparison of clinical results (Outcome Measure 1). Behavioral outcomes were not collected for this historical population and this cohort is not included in the analysis of this outcome measure.
  Ten of the treated subjects in the interventional group did not consent to participate in the biobehavioral phase of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Number analyzed (Participants) | 25 | 0 | 29
units on a scale
  Baseline | 34.8 (8.8) |  | 38.9 (13.0)
  Day 28: number analyzed (Participants) | 22 | 0 | 26
  Day 28 | 42.7 (10.2) |  | 40.3 (12.1)
  Day 100: number analyzed (Participants) | 20 | 0 | 26
  Day 100 | 39.5 (9.1) |  | 40.4 (14.1)
  Day 180: number analyzed (Participants) | 12 | 0 | 21
  Day 180 | 38.6 (9.9) |  | 38.9 (13.4)
Statistical Analysis 1: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Baseline; Test type: Superiority; p = 0.95, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 28; Test type: Superiority; p = 0.26, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 100; Test type: Superiority; p = 0.63, t-test, 2 sided
Statistical Analysis 4: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 180; Test type: Superiority; p = 0.76, t-test, 2 sided

3. Secondary Outcome: Score of Anxiety Symptoms Using the Inventory of Depression and Anxiety Symptoms (IDAS) Instrument
Description: Levels of anxiety symptoms will be measured using the Inventory of Depression and Anxiety Symptoms (IDAS) instrument. (see Watson, 2007). Anxiety will be assessed combining two domain categories of the IDAS (panic and traumatic intrusions). There are seven 5-item, Likert-style questions responding symptom severity "during the past 2 weeks, including today ..." ranging from 'Not at all' to 'Extremely.' Scores range from 0 to 28 with higher scores indicating worse symptoms.
Time Frame: Baseline, Day 28, Day 100 and Day 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Number analyzed (Participants) | 25 | 0 | 29
units on a scale
  Baseline: number analyzed (Participants) | 25 | 0 | 28
  Baseline | 16.0 (5.19) |  | 15.6 (4.5)
  Day 28: number analyzed (Participants) | 21 | 0 | 26
  Day 28 | 17.5 (4.3) |  | 16.9 (4.6)
  Day 100: number analyzed (Participants) | 18 | 0 | 27
  Day 100 | 19.2 (6.0) |  | 17.4 (4.2)
  Day 180: number analyzed (Participants) | 12 | 0 | 21
  Day 180 | 18.6 (6.6) |  | 16.9 (4.7)
Statistical Analysis 1: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Baseline; Test type: Superiority; p = 0.99, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 28; Test type: Superiority; p = 0.48, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Test type: Superiority; p = 0.35, t-test, 2 sided
Statistical Analysis 4: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 180; Test type: Superiority; p = 0.96, t-test, 2 sided

4. Secondary Outcome: Score of Fatigue Symptoms Using the Fatigue Symptom Inventory (FSI) Instrument
Description: Levels of fatigue symptoms will be measured using the Fatigue Symptom Inventory instrument. The FSI comprises 13 eleven-item Likert-style questions ranging from 0 = "Not at all fatigued" to 10 -"Extreme fatigue". The FSI score is the average of the individual question scores. The range of scores is 0 to 10 with higher scores indicate greater fatigue (Hann, 1998).
Time Frame: Baseline, Day 28, Day 100 and Day 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Number analyzed (Participants) | 25 | 0 | 29
units on a scale
  Baseline: number analyzed (Participants) | 25 | 0 | 28
  Baseline | 2.4 (1.5) |  | 4.1 (2.1)
  Day 28: number analyzed (Participants) | 21 | 0 | 26
  Day 28 | 4.2 (1.8) |  | 4.5 (1.6)
  Day 100: number analyzed (Participants) | 20 | 0 | 27
  Day 100 | 3.7 (2.0) |  | 4.3 (1.9)
  Day 180: number analyzed (Participants) | 12 | 0 | 12
  Day 180 | 4.2 (1.1) |  | 4.2 (1.6)
Statistical Analysis 1: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 28; Test type: Superiority; p = 0.75, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 100; Test type: Superiority; p = 0.28, t-test, 2 sided
Statistical Analysis 4: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 180; Test type: Superiority; p = 0.82, t-test, 2 sided

5. Secondary Outcome: Score of Sleep Symptoms Using the Pittsburgh Sleep Quality Index (PSQI) Instrument
Description: Levels of sleep symptoms will be measured using the Pittsburgh Sleep Quality Index instrument. The PSQI contains 19 four-item Likert-style questions conducted over a 30-day period and 5 questions rated by the bed partner or roommate. Responses range from 0 = Not in the past month to 3 = Three or more times a week. The bed partner/roommate questions were not assessed. The 19 self-rated questions are grouped into seven component domains including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. See Buysse (1989), for the scoring schema of the component domains. The PSQI score is the sum of the seven component scores and ranges from 0 to 21. Higher scores indicate poorer sleep quality.
Time Frame: Baseline, Day 28, Day 100 and Day 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Number analyzed (Participants) | 25 | 0 | 29
units on a scale
  Baseline: number analyzed (Participants) | 25 | 0 | 28
  Baseline | 7.5 (4.2) |  | 6.9 (3.9)
  Day 28: number analyzed (Participants) | 21 | 0 | 26
  Day 28 | 8.1 (4.4) |  | 7.8 (4.7)
  Day 100: number analyzed (Participants) | 20 | 0 | 27
  Day 100 | 7.9 (4.5) |  | 6.7 (3.6)
  Day 180: number analyzed (Participants) | 12 | 0 | 21
  Day 180 | 8.5 (4.0) |  | 7.2 (3.9)
Statistical Analysis 1: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Baseline; Test type: Superiority; p = 0.54, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 28; Test type: Superiority; p = 0.61, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 100; Test type: Superiority; p = 0.42, t-test, 2 sided
Statistical Analysis 4: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 180; Test type: Superiority; p = 0.38, t-test, 2 sided

6. Secondary Outcome: Score of Pain Symptoms Using the Brief Pain Inventory (BPI) Instrument (Interference)
Description: Levels of interference in activities due to pain symptoms will be measured using the Brief Pain Inventory (BPI) instrument. The BPI Interference scale is a mean of 7 eleven-item Likert-style questions with a range of 0-10 (0 = Does not interfere to 10 = Completely interferes). Higher scores indicate greater interference in daily activities due to pain symptoms (see Cleeland 1994).
Time Frame: Baseline, Day 28, Day 100 and Day 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) | Historical Control Arm (Primary Outcome Measure) | Historical Control Arm (Secondary Outcome Measures)
Number analyzed (Participants) | 25 | 0 | 29
units on a scale
  Baseline | 1.5 (1.7) |  | 1.8 (2.1)
  Day 28: number analyzed (Participants) | 21 | 0 | 26
  Day 28 | 2.0 (2.0) |  | 1.7 (2.2)
  Day 100: number analyzed (Participants) | 18 | 0 | 27
  Day 100 | 1.6 (1.8) |  | 2.2 (2.7)
  Day 180: number analyzed (Participants) | 12 | 0 | 21
  Day 180 | 1.6 (2.4) |  | 2.3 (2.4)
Statistical Analysis 1: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Baseline; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 28; Test type: Superiority; p = 0.32, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 100; Test type: Superiority; p = 0.63, t-test, 2 sided
Statistical Analysis 4: Comparison: Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) vs Historical Control Arm (Secondary Outcome Measures); Comparison at Day 180; Test type: Superiority; p = 0.30, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events information was not collected for the historical control groups.
Groups:
- Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc): Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant. Methotrexate will be dosed at 15 mg/m2 Day +1 and 10mg/m2 Days +3, +6 and +11. Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1
  Tacrolimus: Patients enrolled in the clinical trial will receive tacrolimus per institutional guidelines at doses to maintain therapeutic levels and continued until at least Day 90 posttransplant.
  Methotrexate: Methotrexate will be dosed at 15 mg/m2 Day +1 and 10mg/m^2 Days +3, +6 and +11.
  Tocilizumab: Tocilizumab will be administered intravenously at a dose of 8 mg/kg at Day -1.
  The adverse events reported (serious and non-serious) include only those events experienced by subjects enrolled at the Medical College of Wisconsin site. Adverse events and serious adverse events were not abstracted from the databases for the two historical control populations.
Arm/Group | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc)
All-Cause Mortality (participants affected / at risk) | 13/35
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) (N=35)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus, Methotrexate and Tocilizumab (Tac/MTX/Toc) (N=35)
Anemia (Blood and lymphatic system disorders) | 23 (23)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 27 (27)
Sepsis (Infections and infestations) | 7 (7)
Alanine aminotransferase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (16)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT02206035/Prot_SAP_002.pdf
  • Informed Consent Form (2015-01-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT02206035/ICF_003.pdf